CLINICAL TRIAL: NCT00826930
Title: Open-label Study to Determine the Effect of Trans Sodium Crocetinate (TSC) on Intra-tumoral Oxygen Concentration, Tolerability, and Pharmacokinetics of TSC in Post-operative Patients With High Grade Glioma (HGG)
Brief Title: Trans Sodium Crocetinate (TSC) Study of Intra-tumoral Oxygen Concentration, Safety, and Pharmacokinetics in Patients With High Grade Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor business decision, not based on safety or efficacy data.
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Responsible Party: Kim M. Whitten, PharmD, RAC, Diffusion Pharmaceuticals LLC
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DP100-201
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: High Grade Glioma
Keywords: High Grade Glioma; Brain Tumor; Solid Tumor; Partial Debulking; Tumor Resection; Tumor Tissue Hypoxia; Radiation Sensitizer; Cancerous Tumor
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — trans-sodium crocetinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1A (Experimental): 0.5 mg/kg TSC, anticonvulsants at Baseline - phenytoin only or none
  Interventions: Drug: Trans Sodium Crocetinate (TSC)
- 2A (Experimental): 0.75 mg/kg TSC, anticonvulsants at Baseline - phenytoin only or none
  Interventions: Drug: Trans Sodium Crocetinate (TSC)
- 3A (Experimental): 1.0 mg/kg TSC, anticonvulsants at Baseline - phenytoin only or none
  Interventions: Drug: Trans Sodium Crocetinate (TSC)
- 4A (Experimental): Dose of TSC either 0.5 mg/kg, 0.75 mg/kg, or 1.0 mg/kg based on the Data Monitoring Committee decision, anticonvulsants at Baseline - phenytoin only or none
  Interventions: Drug: Trans Sodium Crocetinate (TSC)
- 1B (Experimental): 0.5 mg/kg TSC, anticonvulsants at Baseline - any except phenytoin-only or none
  Interventions: Drug: Trans Sodium Crocetinate (TSC)
- 2B (Experimental): 0.75 mg/kg TSC, anticonvulsants at Baseline - any except phenytoin-only or none
  Interventions: Drug: Trans Sodium Crocetinate (TSC)
- 3B (Experimental): 1.0 mg/kg TSC, anticonvulsants at Baseline - any except phenytoin-only or none
  Interventions: Drug: Trans Sodium Crocetinate (TSC)
- 4B (Experimental): Dose of TSC either 0.5 mg/kg, 0.75 mg/kg, or 1.0 mg/kg based on the Data Monitoring Committee decision, anticonvulsants at Baseline - any except phenytoin-only or none
  Interventions: Drug: Trans Sodium Crocetinate (TSC)

INTERVENTIONS:
Drug: Trans Sodium Crocetinate (TSC) — Single bolus intravenous administration in a superficial vein of the arm over a period of up to 2 minutes.

SUMMARY:
The purpose of this study is to evaluate the impact of Trans Sodium Crocetinate (TSC) on oxygen levels in brain tumor tissue in patients with high grade glioma. The proposed clinical indication for TSC is a radiation sensitizer for the treatment of cancerous tumors.

DETAILED DESCRIPTION:
In this open-label, one-site study, up to 48 patients with high grade glioma (HGG) who are undergoing biopsy or partial debulking of the tumor as part of standard of care will have an oxygen monitoring probe placed in residual tumor tissue. Oxygen levels in the tumor tissue will be measured prior to and after administering a single bolus injection of TSC. Safety assessments will occur throughout the trial, including at a 7 to 14 day follow-up visit. Pharmacokinetic assessments will be performed prior to and during the first 24 hours after TSC dosing.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Prior histological diagnosis of high grade glioma (HGG) with prior initial treatment and radiation therapy for HGG; recurrence of HGG suspected, and care plan includes surgical procedure.
* Undergoing surgical procedure for clinical reasons, and gross surgical resection not expected.
* Neurosurgeon is planning stereotactic biopsy or tumor debulking for clinical reasons; frozen tissue confirmation of malignancy during this operative procedure is necessary.
* Neurosurgeon evaluates that placement of oxygen monitoring probe after biopsy or debulking can be done safely without complications.
* Contrast enhancing disease on MRI within 21 days prior to enrollment.
* Karnofsky Performance Score ≥ 60 at Screening.
* Recovered from toxicity of prior antineoplastic therapy, and off cytotoxic chemotherapy for 7 days prior to Screening.
* Recovered from prior radiotherapy and had at least 21 days elapse since completion of radiotherapy prior to Screening.
* Recovered from prior surgery for their brain tumor in investigator's clinical judgment.
* If female, negative serum or urine pregnancy test at Screening.
* Within 2 weeks of starting study, hematologic and renal functions as specified: Absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 9.0g/dL, creatinine ≤ 1.7mg/dl, serum bilirubin ≤ 1.5mg/dL, blood urea nitrogen within 2 times the upper limit of normal, transaminases ≤ 4 times above the upper limits of the institutional norm, and prothrombin time and partial thromboplastin time within institutional norm or below.
* Patient or patient's medical power of attorney provided written consent to participate in the study.
* Mini Mental Status Exam score ≥ 15.

Exclusion Criteria:

* Pregnant or lactating.
* Receiving concurrent cytotoxic chemotherapy for their tumor within 7 days prior to Screening, or decision is made at the time of surgery to treat with other modality of treatment (e.g., gliadel wafers).
* Serious concurrent infection or medical illness which would jeopardize the ability of the patient to safely participate.
* Behavioral, cognitive, or psychiatric disease or personal situation that might interfere with optimal participation.
* Cannot undergo an MRI.
* Received an investigational drug not approved for human use by the FDA within 30 days of enrollment.
* Previously received TSC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in tumor tissue oxygen monitoring recordings | Daily while inpatient
Safety assessments (laboratory tests) | Daily while inpatient, 7-14 Day Follow-up

SECONDARY OUTCOMES:
Pharmacokinetic assessments | Day 1, Day 2
Tumor hypoxia biomarkers (HIF 1-alpha, osteopontin, carbonic anhydrase IX) | Daily while inpatient

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Medical Institute/Johns Hopkins Hospital, Baltimore, Maryland, United States